CLINICAL TRIAL: NCT00458198
Title: Integrated Behavioral Treatment for Selective Mutism
Brief Title: Integrated Behavioral Therapy for Treating Children With Selective Mutism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R34MH070938 (NIH); R34MH070938 (NIH); DDTR B3-PDX
Record Dates: First submitted 2007-04-05; First posted 2007-04-09 (Estimated); Last update posted 2016-11-28 (Estimated); Status verified 2016-11

CONDITIONS: Selective Mutism
Keywords: Selective Mutism
MeSH Terms: conditions — Mutism

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- 1 (Experimental): Participants will receive integrated behavioral therapy
  Interventions: Behavioral: Integrated behavioral therapy (BT)
- 2 (Active Comparator): Participants will receive integrated behavioral therapy after a 12-week waitlist period
  Interventions: Behavioral: Integrated behavioral therapy (BT)

INTERVENTIONS:
Behavioral: Integrated behavioral therapy (BT) — Participants in the BT condition will receive twenty 60-minute sessions over 24 weeks. Sessions will focus on graduated exposure to new speaking situations as the primary agent of anxiety reduction. Behavioral procedures will include systematic desensitization, shaping, and self-modeling procedures. Although a variety of exposure exercises will be routinely conducted in-session, any behavioral assignments will take place outside of session. Behavioral exercises will be implemented, as needed, in a modular fashion. For example, exercises may focus on speaking in-session to therapist, either at school or at home with others present. The therapist will be primarily responsible for developing the exposure parameters, but collaboration of parent, teacher, child will be emphasized increasingly over time. Reinforcement for attempts to complete assignments (contingency management program) will occur throughout treatment.

SUMMARY:
This study will determine the effectiveness of integrated behavior therapy in treating children with selective mutism.

DETAILED DESCRIPTION:
Selective mutism (SM) is a childhood behavior disorder that interferes with social and educational development. It is characterized by a persistent failure to speak in specific social situations, despite being able to speak in other situations. Children with SM typically speak when they are at home with immediate family, but fail to speak in other settings. Behavior therapy (BT), commonly used for treating anxiety disorders and phobias, is a type of treatment that uses training and desensitization methods to help patients become more comfortable in situations that cause anxiety. Based on available evidence, integrated BT, which involves parents, teachers, and the therapist, may be an effective treatment for SM. This study will determine the effectiveness of integrated BT in treating children with selective mutism.

Following a diagnostic assessment to determine eligibility, participants in this single-blind study will be randomly assigned to receive BT either immediately upon study entry or after a 3-month waiting period. BT will consist of 20 1-hour treatment sessions over 6 months. In BT, children will practice speaking to people with whom it has been difficult to speak in the past. Parents, teachers, and children will be taught about anxiety related to SM, setting treatment goals, monitoring anxiety, learning skills to relax, and gradually entering situations that may trigger anxiety. These skills will be practiced during treatment sessions, in school with other children and teachers, and at home on a daily basis. Both parents and teachers will record activities that children have been able to accomplish. In addition, participants will attend study visits at Weeks 8, 12, and 24 for assessments of outcomes.

Participants who are assigned to the waitlist group will not receive treatment during their first 3 months in the study. They will attend study visits at Weeks 8 and 12 to assess any improvement in symptoms. Participants whose symptoms do not improve by the end of the 3-month period may either stop participation or receive 6 months of BT.

All participants will attend one 2- to 3-hour follow-up visit 3 months post-treatment. This visit will include interviews and questionnaires about SM symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of selective mutism
* Score of less than 60 on the Childrens Global Assessment Scale (CGAS)
* Has lived continuously with a primary caretaker who has known the child well for at least 6 months prior to study entry and is legally able to sign the consent form

Exclusion Criteria:

* Diagnosis of any of the following psychiatric disorders: bipolar disorder, pervasive developmental disorder (e.g., Asperger's, autism), mental retardation, or psychotic disorder
* Possibility that a communication disorder may account for the selective mutism
* Current use of or a clinical indication for use of psychotropic medication (youth entering study on a stable psychostimulant regimen for ADHD will not be excluded)
* History of unsuccessful treatment with cognitive behavioral therapy for anxiety that occurred within 2 years prior to study entry
* Any major neurological disorder or major medical illness that may prevent study participation
* Child and/or parent is not English-speaking and is unable to complete measures or treatment without the assistance of a dedicated translator
* Child is not currently attending school (including pre-school), day camp, or other structured daily activity, or has missed more than 50% of school days in the 2 months prior to study entry
* Child's primary teacher is unwilling or unable to participate in the treatment plan

Ages: 4 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 21 (Actual)
Dates: Start 2006-01; Primary Completion 2008-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Selective Mutism Questionnaire | Measured at Weeks 8, 12, 24, and 36
Anxiety Disorders Interview Schedule (ADIS) Severity Rating | Measured at Weeks 8, 12, 24, and 36
Clinical Global Impression | Measured at Weeks 8, 12, 24, and 36

SECONDARY OUTCOMES:
Strong Narrative Assessment Procedure | Measured at Weeks 8, 12, 24, and 36

CONTACTS AND LOCATIONS:
Overall Officials: R. Lindsey Bergman, PhD, Principal Investigator — Semel Institute for Neuroscience & Human Behavior, Univeristy of California Los Angeles (UCLA)
Locations (1):
- 300 UCLA Medical Plaza, Los Angeles, California, United States

REFERENCES:
- [Result] Bergman RL, Gonzalez A, Piacentini J, Keller ML. Integrated Behavior Therapy for Selective Mutism: a randomized controlled pilot study. Behav Res Ther. 2013 Oct;51(10):680-9. doi: 10.1016/j.brat.2013.07.003. Epub 2013 Jul 16. PMID 23933108